CLINICAL TRIAL: NCT01540344
Title: Multimodality Treatment Including Pre- and Postoperative Systemic Chemotherapy Plus Cetuximab, Cytoreductive Surgery (CRS) and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients With Peritoneal Carcinomatosis Arising From Wild Type K-ras Colon Cancer: A Prospective Multicenter Phase II Study.
Brief Title: Combined Anticancer Treatment of Advanced Colon Cancer
Acronym: COMBATAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment.
Sponsor: University of Regensburg (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Pompiliu Piso, Prof. MD, Principal Investigator, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/06/2009; 2009-014040-11 (EudraCT Number)
Record Dates: First submitted 2012-02-19; First posted 2012-02-28 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Peritoneal Carcinomatosis; Colorectal Cancer Metastatic
Keywords: peritoneal carcinomatosis; cytoreductive surgery; HIPEC; colorectal cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): 1. FOLFOX/FOLFIRI + cetuximab (6 cycles)
  2. CRS and HIPEC
  3. FOLFOX/FOLFIRI + cetuximab (6 cycles)
  Interventions: Procedure: CRS; Drug: HIPEC

INTERVENTIONS:
Procedure: CRS — complete macroscopic cytoreduction (CC-0/1)
  Other Names: Cytoreductive surgery
Drug: HIPEC — bidirectional hyperthermic intraperitoneal chemotherapy (HIPEC) with 400 mg/sqm 5-FU + 20 mg/sqm folinic acid IV and 300 mg/sqm oxaliplatin IP
  Other Names: Hyperthermic intraperitoneal chemotherapy

SUMMARY:
The COMBATAC study evaluates the the effect as assessed by progression-free survival (PFS) of perioperative systemic chemotherapy including cetuximab and cytoreductive surgery (CRS) and bidirectional hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with peritoneal carcinomatosis arising from colorectal cancer.

DETAILED DESCRIPTION:
More than 10% of patients with colorectal cancer (CRC) already show peritoneal carcinomatosis at the time of initial diagnosis and up to 25% of all patients develop peritoneal carcinomatosis during the natural course of their disease as a common sign of tumor progression or recurrence.

The existing data suggests that CRS and HIPEC as an integral part of a multidisciplinary treatment concept may improve long-term survival of selected patients with peritoneal carcinomatosis of colonic origin. Moreover, hyperthermic peritoneal perfusion with oxaliplatin in combination with synchronous application of 5-FU/leucovorin seems to improve the efficacy of HIPEC in comparison to a mitomycin C-based intraperitoneal treatment regimen and may lead to a better local tumor control. The improved systemic treatment strategy with neoadjuvant chemotherapy may lead to increased rates of complete macroscopic cytoreduction and together with the adjuvant treatment to better control of distant metastasis and tumor recurrence. However, there is no prospective study available evaluating the clinical and oncological outcome after standard-of-care chemotherapy including targeted anticancer therapy in combination with CRS and HIPEC. The published morbidity and mortality rates after CRS and HIPEC are comparable to other major gastrointestinal surgery and seem to be acceptable considering the expected improvement of oncological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Synchronous or metachronous peritoneal carcinomatosis arising from histologically proven colorectal or appendiceal adenocarcinoma
* Complete macroscopic cytoreduction (CCR-0/1)
* Free treatment interval of at least 6 month after the last chemotherapy
* Age over 18 and below 71 years
* Good general health status (Karnofsky > 70%, ECOG 0-2)
* Absence of hematogenous metastasis (lung, bone, brain, > 3 peripheric resectable liver metastases)
* Absence of contraindication for systemic chemotherapy and/or extended surgery
* Life expectancy greater than 6 months
* Written informed consent
* Creatinine clearance > 50 ml/min, serum creatinine ≤ 1.5 x ULN
* Serum bilirubin ≤ 1.5 x ULN (upper limit of normal), ASAT and ALAT ≤ 2.5 x ULN
* Platelet count > 100,000 /ml, haemoglobin > 9 g/dl, neutrophile granulocytes ≥ 1,500 /ml, International Normalized Ration (INR) ≤ 2
* Absence of peripheral neuropathy > grade 1 (CTCAE v4.0)
* No pregnancy or breast feeding. Adequate contraception in fertile patients.

Exclusion Criteria:

* Incomplete cytoreduction
* Hematogenous metastasis including irresectable liver metastasis
* Prior chemotherapy or therapy with EGFR receptor antibody for metastatic disease
* K-ras mutation
* Known allergy to murine or chimeric monoclonal antibodies
* Histology of signet ring carcinoma
* Other malignancy than disease under study / second cancer
* Impaired liver, renal or hematologic function as mentioned above (inclusion criteria)
* Heart failure NYHA ≥ 2 or significant Coronary Artery Disease
* Alcohol and/or drug abuse
* Patients unable or unwilling to comply with the study protocol, treatment or follow-up
* Patients included in other clinical trials interfering with the present study

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 24 months

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
Feasibility of the combined treatment concept | 9 months
  Assessment of tumor progression, AE and SAE during treatment phase leading to modification or end of treatment.
Quality of life (QoL) | 2 years
  assessed by EORTC-QLQ-C30
Pathohistological regression | 16 weeks
  assessed by Dworak grade of regression in histology after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pompiliu Piso, Prof. MD, Principal Investigator — University of Regensburg
Locations (7):
- Germany (7):
  - Charité Campus Mitte, Humboldt-University Berlin, Berlin
  - Cologne-Merheim Medical Center, University Witten/Herdecke, Cologne
  - Medical Center of the Friedrich-Alexander-University Erlangen- Nürnberg, Erlangen
  - University Hospital Regensburg, Regensburg
  - St. John of God Hospital Regensburg, Regensburg
  - University Hospital, University of Tuebingen, Tübingen
  - University Hospital Wuerzburg, Julius-Maximilians University, Würzburg

REFERENCES:
- [Background] Glockzin G, Rochon J, Arnold D, Lang SA, Klebl F, Zeman F, Koller M, Schlitt HJ, Piso P. A prospective multicenter phase II study evaluating multimodality treatment of patients with peritoneal carcinomatosis arising from appendiceal and colorectal cancer: the COMBATAC trial. BMC Cancer. 2013 Feb 7;13:67. doi: 10.1186/1471-2407-13-67. PMID 23391248
- [Result] Glockzin G, Zeman F, Croner RS, Konigsrainer A, Pelz J, Strohlein MA, Rau B, Arnold D, Koller M, Schlitt HJ, Piso P. Perioperative Systemic Chemotherapy, Cytoreductive Surgery, and Hyperthermic Intraperitoneal Chemotherapy in Patients With Colorectal Peritoneal Metastasis: Results of the Prospective Multicenter Phase 2 COMBATAC Trial. Clin Colorectal Cancer. 2018 Dec;17(4):285-296. doi: 10.1016/j.clcc.2018.07.011. Epub 2018 Jul 31. PMID 30131226